CLINICAL TRIAL: NCT04203563
Title: Strong People Strength Training Program: A Community-Based Randomized Trial
Brief Title: Strong People Strength Training Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell University (Other)
Collaborators: Montana State University (Other); Texas A&M University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MG071019
Record Dates: First submitted 2019-10-10; First posted 2019-12-18 (Actual); Last update posted 2020-07-21 (Actual); Status verified 2020-07

CONDITIONS: Heart Diseases; Cardiovascular Diseases; Diabetes; Sedentary Lifestyle; Overweight and Obesity; Depression, Anxiety; Stress; Fatigue
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Diabetes Mellitus; Sedentary Behavior; Overweight; Obesity; Depression; Anxiety Disorders; Fatigue

STUDY DESIGN:
Intervention Model Description: Group 1 participants attend twice weekly progressive strength training classes with CPR certified and Strong People trained educators in fall 2019 for 12 weeks.
  Group 2 participants receive twice weekly progressive strength training classes in January 2020 for 12 weeks. During the first 12 weeks of the study Group 2 participants do not receive these classes. (Delayed)
Masking Description: Randomization to arm follows the baseline assessment visit.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Group 1 participants attend twice weekly progressive strength training classes with CPR certified and Strong People trained educators in fall 2019 for 12 weeks. Intervention Group.
  Interventions: Behavioral: Strong People Strength Training
- Group 2 (Other): Group 2 participants receive twice weekly progressive strength training classes in January 2020 for 12 weeks. Delayed Intervention Group.
  Interventions: Behavioral: Strong People Strength Training

INTERVENTIONS:
Behavioral: Strong People Strength Training — A community-based progressive strength training program

SUMMARY:
The Strong People Strength Training study aims to assess whether a community-based progressive strength training program can improve risk factors for diabetes and heart disease in older rural adults.

DETAILED DESCRIPTION:
This study aims to evaluate the effects of a twice weekly, 12-week progressive strength training program, Strong People Strength Training, on cardiometabolic risk factors in a pragmatic, community-based randomized intervention trial among rural men and women 50 and older. We hypothesize that individuals randomized to the intervention group will demonstrate statistically significant and clinically meaningful improvements in cardiometabolic risk factors as well as physical function, quality of life, and physical activity compared to those randomized to the delayed intervention control group.

ELIGIBILITY:
Inclusion Criteria:

* Age 50 or older
* Willing and able to get health care provider (HCP) authorization if required (PAR-Q answered yes to any question or 70 and older)

Exclusion Criteria:

* Strength trained in last 12 months
* Previous enrollment in Strong People
* Enrolled or planning to enroll in lifestyle program
* Cognitive impairment
* Unable to obtain physician authorization

Ages: 50 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 167 (Actual)
Dates: Start 2019-08-20 (Actual); Primary Completion 2019-12-23 (Actual); Study Completion 2019-12-23 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Hemoglobin A1c at 12 Weeks | Baseline and outcome (after 12 weeks)
  The hemoglobin A1c test tells you your average level of blood sugar over the past 2 to 3 months. It's also called HbA1c.
Change from Baseline BMI at 12 Weeks | Baseline and outcome (after 12 weeks)
  Body mass index (BMI) is a measure of body fat based on height and weight that applies to adult men and women.
Change from Baseline Weight at 12 Weeks | Baseline and outcome (after 12 weeks)
  body weight
Change from Baseline in American Heart Association's Life's Simple 7 score at 12 Weeks | Baseline and outcome (after 12 weeks)
  The American Heart Association's Life's Simple 7 score is comprised of seven cardiovascular disease (CVD) risk factors: physical activity, healthy diet score, blood glucose, BMI, blood cholesterol, blood pressure, and smoking; each risk factor is categorized as ideal, intermediate, or poor.
  Minimum value is 0, Maximum value is 14. Higher scores on the scale represent a better outcome.

SECONDARY OUTCOMES:
Change from Baseline Cholesterol at 12 Weeks | Baseline and outcome (after 12 weeks)
  Total cholesterol measured with the Alere Cholestech LDX Analyzer
Change from Baseline Resting Heart Rate at 12 Weeks | Baseline and outcome (after 12 weeks)
  Heart rate (beats per minute) while at rest
Change from Baseline Blood Pressure at 12 Weeks | Baseline and outcome (after 12 weeks)
  Blood pressure measured at rest; systolic over diastolic (mm Hg)
Change from Baseline Functional Fitness Tests at 12 Weeks | Baseline and outcome (after 12 weeks)
  Six domains of the functional fitness/ senior fitness tests
Change from Baseline Physical Activity at 12 Weeks measured using accelerometry | Baseline and outcome (after 12 weeks)
  Objective physical activity measured using an accelerometer worn for 7 days
Change from Baseline Physical Activity at 12 Weeks measured using self-report | Baseline and outcome (after 12 weeks)
  Self-report physical activity measured using CHAMPS Activities Questionnaire for Older Adults.
  Questionnaire includes 41 activity questions and participant reports on number of hours per week involved in each activity using possible responses: less than 1 hour; 1-2.5 hours; 3-4.5 hours; 5-6.5 hours; 7-8.5 hours; 9 or more hours. More hours reported corresponds with more time in physical activity.
Change from Baseline Fatigue at 12 Weeks | Baseline and outcome (after 12 weeks)
  Measured with self report using the Visual Analogue Scale to Evaluate Fatigue Severity (VAS-F). This validated scale consists of 18 items relating to the experience of fatigue. Each item the participant responds on a scale of 0 to 10. For example with 0 being not at all tired and 10 being extremely tired.
Change from Baseline Depression using the Center for Epidemiologic Studies Depression Scale (CES-D) at 12 Weeks | Baseline and outcome (after 12 weeks)
  Measured with self report using the Center for Epidemiologic Studies Depression Scale (CES-D). Score ranges from 0 to 60 with with higher scores indicating the presence of more depression symptoms.
Change from Baseline Depression using the Patient Health Questionnaire (PHQ-8) at 12 Weeks | Baseline and outcome (after 12 weeks)
  Measured with self report using the Patient Health Questionnaire (PHQ-8). Score ranges from 0 to 24 with greater scores reflecting more depression symptoms.
Change from Baseline Anxiety at 12 Weeks using the Beck Anxiety Inventory | Baseline and outcome (after 12 weeks)
  Anxiety measured by questionnaire using the Beck Anxiety Inventory which is a 21-question multiple-choice self-report inventory that is used for measuring the severity of anxiety. Scores range from 0 to 63 with higher scores indicating more anxiety.
Change from Baseline Anxiety at 12 Weeks using the the General Anxiety Disorder Scale (GAD-7) | Baseline and outcome (after 12 weeks)
  Anxiety measured by questionnaire using the General Anxiety Disorder Scale (GAD-7) which consists of 7 questions with responses from Not at all, Several Days, More than half hte days, and Nearly every day. Scores range from 0 to 21 with higher scores reflecting more anxiety.
Change from Baseline Stress at 12 Weeks | Baseline and outcome (after 12 weeks)
  Measured with self report using the Perceived Stress Scale (PSS). Scores range from 0 to 40 with higher scores reflecting more perceived stress.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca A Seguin-Fowler, PhD, Principal Investigator — Texas A&M AgriLife Research
Locations (6):
- United States (6):
  - Teton County, Choteau, Montana
  - Chouteau County, Fort Benton, Montana
  - Valley County, Glasgow, Montana
  - Big Horn County, Hardin, Montana
  - Hill County, Havre, Montana
  - Wibaux County, Wibaux, Montana